CLINICAL TRIAL: NCT03434847
Title: The PPREOPP Study: Providing Patients Realistic Expectations of Postoperative Pain
Brief Title: Providing Patients Realistic Expectations of Postoperative Pain
Acronym: PPREOPP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: CMS questions to assess patient satisfaction of pain control were removed from the HCAHPS survey, leaving the study without intervention assessment.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 201709172
Record Dates: First submitted 2017-12-14; First posted 2018-02-15 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, single-blind study
Who Masked: Participant
Masking Description: At enrollment, each patient will be assigned a study number, which will match a previously prepared computer-generated list of randomization numbers to determine whether they will be in the intervention or control arm. Pre-operatively, all patients will complete an initial questionnaire. The patients in the intervention group (n=50) will, in addition to the standard pre-operative assessment, also receive pre-operative educational instruction of what to expect from a post-operative pain perspective including education material to take home.
  For this study, we will be using deception, with the reasoning that the patients' knowledge of the different education materials will affect their rating of the impact of the intervention on satisfaction scores.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard preoperative assessment
- Education (Active Comparator): Pre-operative education regarding post-operative pain expectations
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — Participants who receive perioperative educational to address their expectation about their postoperative pain will have improved pain-related postoperative outcomes.
  Arms: Education

SUMMARY:
Prospective, randomized, single-blind study, whether perioperative educational improves pain-related postoperative outcomes,

DETAILED DESCRIPTION:
This is a prospective, randomized, single-blind study in 100 patients undergoing open colorectal surgery. If the hypothesis is confirmed, then patients who receive perioperative educational interventions to address their expectation about their postoperative pain will have improved pain-related postoperative outcomes.

Randomization and Blinding 100 eligible patients scheduled to undergo open colorectal surgery will be approached in the Center for Preoperative Assessment and Planning Clinic. At enrollment, each patient will be assigned a study number, which will match a previously prepared computer-generated list of randomization numbers to determine whether they will be in the intervention or control arm. Pre-operatively, all patients will complete an initial questionnaire. The patients in the intervention group (n=50) will, in addition to the standard pre-operative assessment, also receive pre-operative educational instruction of what to expect from a post-operative pain perspective including education material to take home.

For this study, deception will be used, with the reasoning that the patients' knowledge of the different education materials will affect their rating of the impact of the intervention on satisfaction scores.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Undergoing open colorectal surgery Able to understand and sign and informed consent form

Exclusion Criteria:

* Age < 18 years
* Unable to complete post-operative CMS questionnaire
* Inability to understand the English language Absolute contraindication to epidural placement (patient refusal, requiring resumption of therapeutic anticoagulation after surgery, anaphylaxis to local anesthetics, local or systemic infections, bleeding diathesis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-10-21 (Actual); Primary Completion 2018-01-16 (Actual); Study Completion 2018-01-16 (Actual)

PRIMARY OUTCOMES:
Does perioperative education improve satisfaction with postoperative pain control at discharge? | Upon discharge, Day 1 - Day 7
  The satisfaction with postoperative pain control will be assessed using an initial, post-operative and discharge questionnaire of participant's pain level, medications (if any) to manage pain, the affects of that pain management, and participant satisfaction of that pain control.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bottros, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koenen P, Bathis H, Schneider MM, Frohlich M, Bouillon B, Shafizadeh S. How do we face patients' expectations in joint arthroplasty? Arch Orthop Trauma Surg. 2014 Jul;134(7):925-31. doi: 10.1007/s00402-014-2012-x. Epub 2014 May 24. PMID 24858373
- [Background] Ghomrawi HM, Mancuso CA, Westrich GH, Marx RG, Mushlin AI; Expectations Discordance Study Group. Discordance in TKA expectations between patients and surgeons. Clin Orthop Relat Res. 2013 Jan;471(1):175-80. doi: 10.1007/s11999-012-2484-3. PMID 22821348
- [Background] Waljee J, McGlinn EP, Sears ED, Chung KC. Patient expectations and patient-reported outcomes in surgery: a systematic review. Surgery. 2014 May;155(5):799-808. doi: 10.1016/j.surg.2013.12.015. Epub 2013 Dec 16. PMID 24787107
- [Background] Shuldham C. A review of the impact of pre-operative education on recovery from surgery. Int J Nurs Stud. 1999 Apr;36(2):171-7. doi: 10.1016/s0020-7489(99)00010-3. PMID 10376227
- [Background] Snyder-Ramos SA, Seintsch H, Bottiger BW, Motsch J, Martin E, Bauer M. Patient satisfaction and information gain after the preanesthetic visit: a comparison of face-to-face interview, brochure, and video. Anesth Analg. 2005 Jun;100(6):1753-1758. doi: 10.1213/01.ANE.0000153010.49776.E5. PMID 15920209
- [Background] Kaur H, Singh G, Singh A, Sharda G, Aggarwal S. Evolving with modern technology: Impact of incorporating audiovisual aids in preanesthetic checkup clinics on patient education and anxiety. Anesth Essays Res. 2016 Sep-Dec;10(3):502-507. doi: 10.4103/0259-1162.177187. PMID 27746541
- [Background] Noorian C, Aein F. Comparative investigation of the effectiveness of face-to-face verbal training and educational pamphlets on readiness of patients before undergoing non-emergency surgeries. J Educ Health Promot. 2015 May 19;4:45. doi: 10.4103/2277-9531.157231. eCollection 2015. PMID 26097859
- See also: HCAHPS Patient Level Correlations — http://www.hcahpsonline.org